CLINICAL TRIAL: NCT05808686
Title: Ischemic Conditioning to Promote Microvascular Resiliency in Frail Individuals
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Matthew J. Durand, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00046569
Record Dates: First submitted 2023-03-28; First posted 2023-04-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Aging; Fragility; Endothelial Dysfunction
Keywords: Vasodilation; Exercise; Fitness
MeSH Terms: conditions — Aneurysm; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ischemic Conditioning-Low (Sham Comparator): We will use a randomized block design to randomize individuals into either Ischemic Conditioning-Low or Ischemic Conditioning-High group using an online randomizer. A handheld sphygmomanometer and blood pressure cuff will be given to study participants. For the Ischemic Conditioning-Low group participants, while sitting, the cuff will be placed around the non-dominant upper arm and inflated to 10 mmHg for 5 min, then released for a 5-min recovery period. A 5-min inflation period is most used. Five cycles of inflation/recovery will be performed. All participants will perform the intervention daily for 2 weeks. Participants will complete daily log sheets documenting the time and pressure of each cuff inflation.
  Interventions: Other: Ischemic Conditioning
- Ischemic Conditioning-High (Experimental): We will use a randomized block design to randomize individuals into either Ischemic Conditioning-Low or Ischemic Conditioning-High group using an online randomizer. A handheld sphygmomanometer and blood pressure cuff will be given to study participants. For the Ischemic Conditioning-High group participants, while sitting, the cuff will be placed around the non-dominant upper arm and inflated to 225 mmHg for 5 min, then released for a 5-min recovery period. A 5-min inflation period is most used. Five cycles of inflation/recovery will be performed. All participants will perform the intervention daily for 2 weeks. Participants will complete daily log sheets documenting the time and pressure of each cuff inflation.
  Interventions: Other: Ischemic Conditioning

INTERVENTIONS:
Other: Ischemic Conditioning — We will use a randomized block design to randomize individuals into either Ischemic Conditioning-Low or Ischemic Conditioning-High group using an online randomizer. A handheld sphygmomanometer and blood pressure cuff will be given to study participants. For the Ischemic Conditioning-High group participants, while sitting, the cuff will be placed around the non-dominant upper arm and inflated to 225 mmHg for 5 min, then released for a 5-min recovery period. A 5-min inflation period is most used. Five cycles of inflation/recovery will be performed. For the Ischemic Conditioning-Low group participants, the cuff will be inflated to 10 mmHg instead. All participants will perform the intervention daily for 2 weeks. Participants will complete daily log sheets documenting the time and pressure of each cuff inflation.

SUMMARY:
The goal of this clinical trial is to see how small blood vessels respond to the stress of high intensity exercise, and if a safe and simple intervention called ischemic conditioning can protect blood vessels from the stress of exercise.

Participants will come in for 3 study visits and get home-based ischemic conditioning. At Study Visit 1, participants will be assessed for their frailty and physical function. Afterwards, they will perform an exercise test. At Study Visit 2, patients will undergo 2 microvascular assessments, perform a high-intensity exercise, then undergo the same 2 microvascular assessments again. Participants will be given a handheld sphygmomanometer and a blood pressure cuff to take home. Depending on which group the participants get randomized into, participants will place the blood pressure cuff around their non-dominant upper arm and inflate to either a low or high pressure for 2 weeks at home. Participants will repeat the same steps in Study Visit 2 for Study Visit 3. In addition, participants will also be assessed for their frailty and physical function.

DETAILED DESCRIPTION:
In elderly individuals the small blood vessels that regulate blood flow to organs and other tissues can become damaged when they are exposed to stress, which can lead to complications following stressful events like surgery. In this study we will examine how these blood vessels respond to the stress of high intensity exercise, and if a safe and simple intervention called ischemic conditioning can increase resiliency of these vessels.

Our previous work showed that conditioned athletes are protected from the stress of a single, high intensity exercise bout whereas non-athletes are not. Others have shown that elderly individuals have reduced large artery function following the high intensity exercise. This study will be the first to examine how the small blood vessels respond to this stress in the elderly. Participants will be asked to come in for 3 study visits.

Study Visit 1

1. Complete assessments on frailty and physical function
2. Complete an exercise test using either a total body recumbent stepper or a bicycle and pedal in a seated position

Study Visit 2

1. Undergo a blood draw to measure plasma sphingolipids
2. Have a CytoCam device take images of small vessels inside their mouth
3. Be assessed by the Laser Doppler Flowmeter while small doses of a vasodilator called acetylcholine are infused into the skin and the local temperature increases
4. Complete a high-intensity interval exercise on a bicycle or an elliptical machine
5. Have a CytoCam device take images of small vessels inside their mouth
6. Be assessed by the Laser Doppler Flowmeter while small doses of a vasodilator called acetylcholine are infused into the skin and the local temperature increases

Home-based Ischemic Conditioning

1. Get a handheld sphygmomanometer and a blood pressure cuff to take home.
2. Depending on which group the participants get randomized into, participants will place blood pressure cuff around non-dominant upper arm and inflate to either a low or high pressure.
3. This intervention will be completed 5 times a day for 2 weeks

Visit 3

1. Undergo a blood draw to measure plasma sphingolipids
2. Have a CytoCam device take images of small vessels inside their mouth
3. Be assessed by the Laser Doppler Flowmeter while small doses of a vasodilator called acetylcholine are infused into the skin and the local temperature increases
4. Complete assessments on frailty and physical function
5. Complete an exercise test using either a total body recumbent stepper or a bicycle and pedal in a seated position
6. Complete a high-intensity interval exercise on a bicycle or an elliptical machine
7. Have a CytoCam device take images of small vessels inside their mouth
8. Be assessed by the Laser Doppler Flowmeter while small doses of a vasodilator called acetylcholine are infused into the skin and the local temperature increases

ELIGIBILITY:
Inclusion Criteria:

* Women and men ages 65-85 years of age

Exclusion Criteria:

* Myocardial infarction in last 6 months
* morbid obesity (BMI >40)
* heart failure
* uncontrolled hypertension
* other condition that precludes high intensity exercise (ex, neurological disorder, acute systemic infection)
* history of blood clots in the extremities
* any condition in which compression of the arm or transient ischemia is contraindicated (e.g., wounds in the arm).

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in Acetylcholine-mediated dilation | 2 hours
  Cutaneous vascular conductance in response to acetylcholine infusion will be calculated as laser Doppler flux / mean arterial pressure
Change in Perfused Vessel Density | 0.5 hours
  Total vessel density (TVD) will be calculated using the DeBacker Score manual analysis on all images that have a minimum microcirculation image quality score (MIQS) of 10. Perfused vessel density (PVD) will be calculated by multiplying total vessel density (TVD) x proportion of perfused vessels (PPV%).

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Wauwatosa, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share individual participant data with other researchers.